CLINICAL TRIAL: NCT00490581
Title: Evaluation of the Housing First Initiative of Chicago Housing for Health Partnership
Brief Title: Evaluation of Housing First Initiative for Chicago Homeless With Chronic Medical Illness
Acronym: CHHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook County Health (Other Government)
Collaborators: Research and Education Foundation of Michael Reese Hospital (Other)
Responsible Party: Principal Investigator, Pamela Gonzalez Sr Director Clinical Research Office, Dir Clinical Research Office, Cook County Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 03-107B JHSH2003-107 IRB
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Unstable Housing
Keywords: Early housing after hospitalization
MeSH Terms: interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): These patients are assigned to the intervention of early supportive housing with case management integrated into the medical system. These subjects are offerred respite care/interim housing upon discharge from enrolling hospitalizations, followed by stable housing within 90 days. They have a case manager at each stage (hospital, respite/interim housing, and stable housing)
  Interventions: Other: case management and supportive housing
- Usual Care (No Intervention): These patients receive usual social services for hospital discharge planning.

INTERVENTIONS:
Other: case management and supportive housing — patients randomized to the study group are offerred respite care/interim housing and case management upon discharge from enrolling hospitalization. They are also offerred stable housing within 90 days of enrolling hospital discharge, with case management at all 3 stages - hospital, respite care/interim housing, and stable housing.
  Arms: Study group

SUMMARY:
The study hypothesizes that early housing after hospitalization with case management integrated into the health and housing systems, will results in decreased use of costly health services (i.e., hospitalizations and Emergency Room visits) with no negative affect on health. To address this hypothesis the investigators implemented a Randomized controlled trial of 407 homeless adults with chronic medical illness in Chicago. Eligible homeless adults were enrolled during a hospitalization to intervention - Early housing with case management - or usual care - usual case management and housing options. The investigators followed the sample for 18 months with assessments at baseline, 1,3,6,9,12 and 18 months are enrollment. Study measures include Quality of Life, Health service use, Alcohol and Substance Use, housing and social and demographic characteristics.

DETAILED DESCRIPTION:
The Chicago Housing for Health Partnership (CHHP) was developed to meet the challenge of providing housing to the most disadvantaged homeless people in the city: those with chronic illnesses who are being discharged from a hospital. The program model was community based and collaboratively created and monitored by an oversight committee composed of the leadership of all involved partner agencies. The CHHP was a group of 8 nonprofit agencies that provided supportive housing and 2 agencies that provided interim housing or respite care. Supportive housing was defined by the intervention as housing without time limits combined with services to help participants to live more stable, productive lives.

To evaluate this new service model, a prospective randomized trial was designed to examine the effect of supportive housing and intensive case management on health service utilization. The investigators enrolled homeless patients with at least 1 of 15 chronic illnesses from 2 urban hospitals that were members of the partnership and known to have large numbers of unstably housed patients. The chronic illnesses were associated with increased mortality in the homeless21 and were verified through review of physician hospital notes. This trial is the health outcomes portion of CHHP.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English or spanish speaking
* Presence of at least one chronic medical illness
* Unstable housing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2003-09; Primary Completion 2007-12 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Hospitalized days - length of stay Emergency Room visits | 18 months
  All days admitted to an inpatient acute care intuition from time of enrollment to study end

CONTACTS AND LOCATIONS:
Overall Officials: laura s sadowski, md, mph, Principal Investigator — Collaborative Research Unit, Stroger Hospital of Cook County
Locations (1):
- John Stroger Hospital of Cook County, Chicago, Illinois, United States

REFERENCES:
- [Derived] Basu A, Kee R, Buchanan D, Sadowski LS. Comparative cost analysis of housing and case management program for chronically ill homeless adults compared to usual care. Health Serv Res. 2012 Feb;47(1 Pt 2):523-43. doi: 10.1111/j.1475-6773.2011.01350.x. Epub 2011 Nov 18. PMID 22098257
- [Derived] Sadowski LS, Kee RA, VanderWeele TJ, Buchanan D. Effect of a housing and case management program on emergency department visits and hospitalizations among chronically ill homeless adults: a randomized trial. JAMA. 2009 May 6;301(17):1771-8. doi: 10.1001/jama.2009.561. PMID 19417194